CLINICAL TRIAL: NCT01553669
Title: The Effects of Reminiscence Therapy on Depression, Self Esteem, Life Satisfaction, and Loneliness of the Elderly in China
Brief Title: Reminiscence Therapy on Depression, Self Esteem, Life Satisfaction, and Loneliness of the Elderly
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese Academy of Sciences (Other Government)
Responsible Party: Principal Investigator, Li Juan, Professor, Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2009BAI77B03
Record Dates: First submitted 2012-03-06; First posted 2012-03-14 (Estimated); Last update posted 2012-05-15 (Estimated); Status verified 2012-05

CONDITIONS: Depression
MeSH Terms: conditions — Depression

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- reminiscence therapy (Experimental): Reminiscence therapy is a method of using the memory to protect mental health and improve the quality of life.
  Interventions: Behavioral: reminiscence therapy
- Control group (No Intervention): The participants assigned to the waiting-list as the control group will be treated as before. After the intervention period, we will conduct reminiscence therapy on them if they ask for.

INTERVENTIONS:
Behavioral: reminiscence therapy — The subjects who are arranged to the experiment group will be intervened using the reminiscence therapy manual proposed by Watt and Cappeliez (2000). According to the manual, the group consisted of six weekly sessions of 90 min each. There will be about four people in each subgroup. During each weekly session, the memories recalled focused on a different theme.
  Other Names: life review
  Arms: reminiscence therapy

SUMMARY:
The primary hypothesis is, comparing with the control group, reminiscence therapy is significantly and clinically effective to improve the experiment group's depressive symptoms after six weeks therapy, and the efficacy can be maintained on the three months follow-up.

The secondary hypothesis is, comparing with the control group, reminiscence therapy significantly reduce the loneliness and increase the self-esteem and life satisfaction of the experiment group.

DETAILED DESCRIPTION:
The subjects who are arranged to the experiment group will be intervened using the reminiscence therapy manual proposed by Watt and Cappeliez (2000). According to the manual, the group consisted of six weekly sessions of 90 min each. During each weekly session, the memories recalled focused on a different theme.

Data collection will occur on screening (as for baseline or pre-test), after intervention immediately (as for post-test), and three months after the intervention (as for follow-up). And outcome measures use standardized instruments with demonstrated validity and reliability:

Geriatric Depression Scale (GDS) Rosenberg self-esteem scale (SES) Life Satisfaction Index A (LSI-A) Russell's UCLA Loneliness Scale

ELIGIBILITY:
Inclusion Criteria:

1. 60 years of age and older;
2. A score above 10 and lower than 26 on the Geriatric Depression Scale (GDS);
3. A score of 24 or higher on the Mini-Mental State Examination (MMSE);
4. Not taking anti-depressant medication or taking part in other psychotherapy when enrolling, if taking anti-depressant medication, must be stabilized on that medication for at least three months;
5. Having no problem with communication (such as, can speak fluent mandarin, or if he/she speaks a dialect, his/her dialect can be understood by most of people).

Exclusion Criteria:

1. Suicide attempt;
2. A diagnosis of cognitive impairment by DSM-Ⅳ, or mental disorders other than depression;
3. Alcohol or drug abuse;
4. Cannot grantee attending the therapy at a weekly base due to physical impairment, lack of time or unwilling etc.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2011-10; Primary Completion 2012-09 (Estimated); Study Completion 2012-09 (Estimated)

PRIMARY OUTCOMES:
Change in depression using the Geriatric Depression Scale(GDS) | the 6th and 18th week

SECONDARY OUTCOMES:
Change in self esteem using the Self-Esteem Scale (SES) | the 6th and 18th week
Change in life satisfaction using the Life Satisfaction Index A (LSI-A) | the 6th and 18th week
Change in loneliness using Russell's UCLA Loneliness Scale | the 6th and 18th week

CONTACTS AND LOCATIONS:
Overall Officials: Juan Li, PhD, Principal Investigator — Chinese Acad Sci, Inst Psychol, Ctr Ageing Psychol, Key Lab Mental Hlth
Locations (1):
- Chinese Academy of Sciences, Institute of Psychology, Center on Ageing Psychology, Key Lab of Mental Health, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chen TJ, Li HJ, Li J. The effects of reminiscence therapy on depressive symptoms of Chinese elderly: study protocol of a randomized controlled trial. BMC Psychiatry. 2012 Nov 5;12:189. doi: 10.1186/1471-244X-12-189. PMID 23126676